CLINICAL TRIAL: NCT03708029
Title: A Clinical Investigation Into the Efficacy of Full-thickness Human Placental Graft (Revita) in Diabetic Foot Ulcers
Brief Title: Efficacy of Human Placental Graft in Diabetic Foot Ulcers
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low enrollment.
Sponsor: StimLabs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SLRV-POD-WC-001
Record Dates: First submitted 2018-10-12; First posted 2018-10-16 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Diabetic Foot
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Treatment (Experimental): Will receive Revita allograft for wound treatment
  Interventions: Other: Revita Allograft
- Control (No Intervention): Will receive current standard of care for wound treatment

INTERVENTIONS:
Other: Revita Allograft — Human placental allograft
  Arms: Intervention Treatment

SUMMARY:
To determine the efficacy of full-thickness placental allograft in chronic wound healing

DETAILED DESCRIPTION:
To evaluate the efficacy of Revita full thickness placental allograft in improving wound closure rates and mean closure time in diabetic foot ulcers (DFUs) as compared to the current standards of wound care treatment

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients
* 18-80 years old
* Diagnosis of Type 1 or 2 Diabetes Mellitus
* Foot ulcers >1cm2 and <25cm2 for 4 weeks or more prior to enrollment
* Able to give consent to participate
* Compliance with all aspects of protocol and follow-up

Exclusion Criteria:

* Male and female patients younger than 18 years old
* Male or female patients older than 80 years old
* Smoking, and any additional health risk factors contraindicated with Revita use
* Involvement in any other ongoing studies

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-11-13 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Complete Wound Closure | 12 weeks
  100% epithelization

SECONDARY OUTCOMES:
Percent(%) Healed | 12 weeks
  Percentage of wound healed

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Research Manager, Study Director — StimLabs
Locations (3):
- United States (3):
  - Gulf Coast Podiatry, Pensacola, Florida
  - Louisiana Foot and Ankle Specialists, Lake Charles, Louisiana
  - Crozer/Keystone Health System, Center for Wound Healing, Springfield, Pennsylvania